CLINICAL TRIAL: NCT00357760
Title: A Randomized Phase II Study to Determine the Effect of 2 Different Doses of AVE0005 (VEGF Trap) in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Ziv-Aflibercept in Treating Patients With Metastatic or Unresectable Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00559; NCI-2009-00559 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E4805 (Other: ECOG-ACRIN Cancer Research Group); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-05

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Metastatic Renal Cell Carcinoma; VEGF Trap
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (higher dose of VEGF Trap) (Experimental): Patients receive a higher dose of ziv-aflibercept (VEGF Trap) IV over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: VEGF Trap
- Arm B (lower dose of VEGF Trap) (Experimental): Patients receive a lower dose of ziv-aflibercept (VEGF Trap) IV over 1 hour on day 1. In both arms, courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. At the time of disease progression, the dose of ziv-aflibercept (VEGF Trap) may be escalated to the higher dose in Arm A.
  Interventions: Biological: VEGF Trap

INTERVENTIONS:
Biological: VEGF Trap — Given IV
  Other Names: AVE0005; Vascular Endothelial Growth Factor Trap; Ziv-Aflibercept

SUMMARY:
This randomized phase II trial studies how well ziv-aflibercept (VEGF Trap) works in treating patients with kidney cancer that has spread from the primary site to other places in the body (metastatic) or is unable to be removed with surgery (unresectable). Ziv-aflibercept may stop the growth of kidney cancer by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of two different doses of AVE0005 (vascular endothelial growth factor [VEGF] Trap [ziv-aflibercept]) treatment on the progression-free proportion at 8 weeks in patients with metastatic renal cell carcinoma who had previous treatment with a tyrosine kinase inhibitor (TKI).

SECONDARY OBJECTIVES:

I. To determine the effect of AVE0005 (VEGF Trap) treatment on objective response rate in patients with metastatic renal cell carcinoma who have had previous TKI treatment.

II. To describe progression-free survival among patients who undergo dose escalation following progression on low-dose AVE0005 (VEGF Trap).

III. To evaluate the safety and tolerability of AVE0005 (VEGF Trap) in patients with metastatic renal cell carcinoma who have had previous treatment with a TKI.

OTHER PRE-SPECIFIED OBJECTIVES:

I. To determine the circulating levels of VEGF AVE0005 (VEGF-Trap) complex and correlate it with clinical activity.

II. To evaluate the modulation of specific angiogenesis-related protein expression by AVE0005 (VEGF Trap).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A (Higher dose of VEGF Trap): Patients receive a higher dose of ziv-aflibercept intervenously (IV) over 1 hour on day 1.

ARM B (Lower dose of VEGF Trap): Patients receive a lower dose of ziv-aflibercept IV over 1 hour on day 1.

In both arms, courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients receiving treatment on Arm B may crossover and receive treatment on Arm A at the time of disease progression.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or unresectable renal cell carcinoma; disease must be conventional clear cell carcinoma or have a component of clear cell carcinoma
* Patient must have measurable lesions according to the Response Evaluation Criteria In Solid Tumors (RECIST); baseline measurements must be performed =< 4 weeks prior to randomization
* Patient must have evidence of progressive disease following treatment with a tyrosine kinase inhibitor (TKI) as assessed by the site investigator on the basis of computed tomography (CT) scans and other appropriate clinical documentation
* Patient must have received at least one prior treatment with a VEGF receptor tyrosine kinase inhibitor for at least 12 weeks; prior treatment with either temsirolimus or everolimus is allowed; prior immunotherapy is limited to cytokine therapy with interleukin 2 and interferon alpha only
* Previous radiotherapy (RT) is permissible provided the measurable disease is outside the RT port; RT must be completed >= 3 weeks prior to randomization
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patient must have recovered from any toxic effects of prior radiotherapy or surgical procedures within 4 weeks prior to randomization
* Adequate organ function as defined in the protocol
* For women of childbearing potential, a negative serum pregnancy test is required within 1 week prior to randomization
* Women of childbearing potential and sexually active males must agree to use an accepted and effective method of contraception while on this study, and for 6 months after the completion of the study; if a woman becomes pregnant while she is on this study or within 6 months after the last dose of protocol therapy, she must inform her treating physician immediately; if a man impregnates a woman while he is on this study or within 6 months after the last dose of protocol therapy, he must inform his treating physician immediately
* Patients who have had basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, ductal carcinoma in situ of the breast, or lobular carcinoma in situ of the breast within the past five years are eligible only if treated with curative intent; patients with other malignancies are eligible only if they have been continuously disease-free for > 5 years prior to the time of randomization

Exclusion Criteria:

* True papillary, sarcomatoid features without any clear cell component, chromophobe, oncocytoma, collecting duct tumors and transitional cell carcinoma are not eligible
* Prior immunotherapy other than cytokine therapy with interleukin 2 and interferon alpha
* Prior treatment with bevacizumab
* Prior cellular therapy, vaccine, hormonal or chemotherapy for renal cell carcinoma; prior therapy for other cancers is allowable if therapy ended at least 5 years prior to enrollment
* History of metastatic central nervous system (CNS) disease
* Pregnant or breastfeeding
* Myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class III or IV congestive heart failure, cerebrovascular accident or transient ischemic attack within 24 weeks prior to randomization
* Prior pulmonary embolism, deep vein thrombosis, or other thromboembolic event
* History of uncontrolled or labile hypertension, with or without antihypertensive drug treatment, within 12 weeks prior to drug administration; this is defined as blood pressure > 150/100 mm Hg or systolic blood pressure > 180 mm Hg on at least 2 repeated determinations on separate days
* Active infection, evidence of bleeding or intratumoral bleeding, or underlying bleeding disorder
* History of hypersensitivity to any Trap agents or recombinant proteins
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pili, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (205):
- United States (204):
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg Cottage Plaza Office, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Nevada Cancer Institute-Summerlin Campus, Las Vegas, Nevada
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - New York Oncology Hematology PC -Albany Medical Center, Albany, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Beth Israel Medical Center, New York, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Scott and White Memorial Hospital, Temple, Texas
  - West Virginia University Charleston, Charleston, West Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 12/21/2007 and closed to accrual on 12/6/2013 with a total accrual of 94 patients.
Period: Overall Study
Arm/Group | Arm A (Higher Dose of VEGF Trap) | Arm B (Lower Dose of VEGF Trap)
Started | 59 | 35
Patients Who Started Treatment | 57 | 34
Eligible and Treated Patients | 57 | 32
Patients Who Undergo Dose Escalation | 0 (Only patients who progressed on the low dose (Arm B) had the opportunity to undergo dose escalation.) | 16
Completed | 0 (Patients continued receiving protocol treatment until progressive disease or unacceptable toxicity.) | 0 (Patients continued receiving protocol treatment until progressive disease or unacceptable toxicity.)
Not Completed | 59 | 35
Not completed — Disease progression | 44 | 17
Not completed — Adverse Event | 10 | 7
Not completed — Death | 0 | 3
Not completed — Alternative therapy | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Never started treatment | 2 | 1
Not completed — Ineligible | 0 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — To receive hospice care | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Higher Dose of VEGF Trap) | Arm B (Lower Dose of VEGF Trap) | Total
Number analyzed (Participants) | 57 | 32 | 89
Age, Continuous [Median (Full Range); unit: years] | 60 [35 to 80] | 62 [33 to 73] | 61 [33 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 43 | 22 | 65

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Alive and Progression-free at 8 Weeks
Description: Progression-free survival (PFS) was defined as time from randomization to the earlier of documentation of progression or death. The proportion of patients who are progression-free and alive at 8 weeks was estimated using the Kaplan-Meier method and the confidence interval was estimated using log transformation method.
  Progression is defined using Response Evaluation Criteria In Solid Tumors (RECIST), as a 20% increase in the sum of the longest diameters of target lesions, or the appearance of new lesions, or unequivocal progression of existing nontarget lesions.
Time Frame: Assessed at 8 weeks
Population: Eligible and treated patients are included in this analysis.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Higher Dose of VEGF Trap) | Arm B (Lower Dose of VEGF Trap)
Number analyzed (Participants) | 57 | 32
proportion of participants | 0.70 [0.59 to 0.79] | 0.52 [0.37 to 0.66]

2. Secondary Outcome: Proportion of Patients With Objective Response
Description: Objective response is defined as complete response (CR) or partial response (PR) determined by Solid Tumor Response Criteria (RECIST).
  CR: The disappearance of all target lesions without the appearance of new lesion(s) and/or unequivocal progression of existing non-target lesions.
  PR: At least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter without the appearance of new lesion(s) and/or unequivocal progression of existing non-target lesions.
  To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no less than four weeks after the criteria for response are first met.
Time Frame: Assessed every 8 weeks while on treatment and then every 3 months until patient is 2 years from enrollment, and then every 6 months until patient is 3 years from enrollment
Population: Eligible and treated patients are included in this analysis.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Higher Dose of VEGF Trap) | Arm B (Lower Dose of VEGF Trap)
Number analyzed (Participants) | 57 | 32
proportion of participants | 0.053 [0.014 to 0.13] | 0.031 [0.002 to 0.14]

3. Secondary Outcome: Progression-free Survival (PFS) Among Patients Who Undergo Dose Escalation Following Progression on Lower-dose VEGF Trap
Description: Patients who progressed on the 1 mg/kg dose (Arm B) at 8 weeks would have the opportunity to receive the 4 mg/kg dose. PFS is defined as the time from dose escalation to disease progression or death, whichever occurs first.
  Disease progression is defined using Response Evaluation Criteria In Solid Tumors (RECIST), as a 20% increase in the sum of the longest diameters of target lesions, or the appearance of new lesions, or unequivocal progression of existing nontarget lesions.
Time Frame: as for outcome 2
Population: Only patients who progressed on the low dose (Arm B) and underwent dose escalation were included in this analysis.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Arm A (Higher Dose of VEGF Trap) | Arm B (Lower Dose of VEGF Trap)
Number analyzed (Participants) | 0 | 16
weeks |  | 14.57 [7.57 to 33.00]

4. Other Pre Specified Outcome: Circulating Levels of VEGF-Trap Complex
Time Frame: Assessed at baseline, 4 weeks, 6 weeks, 8 weeks and end of treatment
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Angiogenesis-related Protein Expression
Time Frame: Assessed every 8 weeks during treatment and end of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 2 weeks while on treatment and for 30 days after the end of treatment, assessed up to 3 years
Arm/Group | Arm A (Higher Dose of VEGF Trap) | Arm B (Lower Dose of VEGF Trap)
Serious Adverse Events (participants affected / at risk) | 35/57 | 18/34
Other Adverse Events (participants affected / at risk) | 52/57 | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Higher Dose of VEGF Trap) (N=57) | Arm B (Lower Dose of VEGF Trap) (N=34)
Anemia (Blood and lymphatic system disorders) | 2 | 3
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Cardiac-ischemia (Cardiac disorders) | 1 | 0
Cardiac troponin I (cTnI) increased (Investigations) | 0 | 1
Hypertension (Vascular disorders) | 20 | 5
Hypotension (Vascular disorders) | 1 | 0
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 2 | 7
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1
CNS, hemorrhage (Nervous system disorders) | 0 | 1
Urinary hemorrhage NOS (Renal and urinary disorders) | 0 | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 9 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 2 | 0
Back, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Head/headache (Nervous system disorders) | 2 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Renal/GU-other (Renal and urinary disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Higher Dose of VEGF Trap) (N=57) | Arm B (Lower Dose of VEGF Trap) (N=34)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Anemia (Blood and lymphatic system disorders) | 11 | 11
Hemolysis (Blood and lymphatic system disorders) | 5 | 0
Leukocytes decreased (Investigations) | 5 | 1
Neutrophils decreased (Investigations) | 2 | 2
Platelets decreased (Investigations) | 5 | 3
Hypertension (Vascular disorders) | 22 | 10
Fatigue (General disorders) | 36 | 24
Fever w/o neutropenia (General disorders) | 1 | 2
Rigors/chills (General disorders) | 0 | 3
Sweating (Skin and subcutaneous tissue disorders) | 2 | 2
Weight loss (Investigations) | 7 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 4 | 2
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 22 | 16
Constipation (Gastrointestinal disorders) | 11 | 10
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 11 | 8
Dry mouth (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 0 | 4
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 5 | 6
Nausea (Gastrointestinal disorders) | 11 | 17
Taste disturbance (Nervous system disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 1 | 6
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Pleura, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Edema limb (General disorders) | 4 | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 2
Alkaline phosphatase increased (Investigations) | 4 | 5
Alanine aminotransferase increased (Investigations) | 6 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2
Creatinine increased (Investigations) | 8 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 4
Proteinuria (Renal and urinary disorders) | 25 | 20
Hyponatremia (Metabolism and nutrition disorders) | 7 | 7
Dizziness (Nervous system disorders) | 5 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Neuropathy-sensory (Nervous system disorders) | 2 | 4
Abdomen, pain (Gastrointestinal disorders) | 0 | 2
Back, pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Chest/thoracic pain NOS (General disorders) | 2 | 3
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Head/headache (Nervous system disorders) | 17 | 8
Joint, pain (Musculoskeletal and connective tissue disorders) | 11 | 8
Muscle, pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Pain-other (General disorders) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 12
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less